CLINICAL TRIAL: NCT03435770
Title: Evaluation of Safety and Feasibility of Endoscopic Ultrasound (EUS)-Guided Radiofrequency Ablation (RFA) for Solid Pancreatic Neoplasms
Brief Title: Evaluation of Safety and Feasibility of EUS-guided RFA for Solid Pancreatic Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Chin Yung Ka, Principal Investigator, Singapore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2702
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms; Pancreatic Adenocarcinoma; Pancreatic Neuroendocrine Tumor; Pancreatic Ductal Adenocarcinoma
Keywords: EUS-guided RFA; Endoscopic ultrasound; radio frequency ablation
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell

STUDY DESIGN:
Intervention Model Description: prospective, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUSRA RFA needle (Experimental): This procedure is very similar to the standard technique of EUS-guided fine needle aspiration. All patients would undergo EUS with a linear array or therapeutic echoendoscope. The location and size of the lesion would be assessed for suitability of treatment. After locating the lesion, the EUSRA RFA needle would be inserted to the centre of the lesion. RFA would then be initiated and hyperechoic interferences would be observed around the electrode signifying heating of the tissue.
  Interventions: Device: EUSRA RFA needle

INTERVENTIONS:
Device: EUSRA RFA needle — A 19-gauge RFA electrode and a RF generator with a electrode that is needle-shaped and echogenic that allows EUS guided puncture of the target lesion. The active electrode tip is 1 cm in length. During ablation, the RF electrode is cooled and perfused internally with circulating chilled saline solution (0°C) delivered via a pump to maintain a constant temperature. A setting of 50W energy would be used for RFA and the duration of application is 10 seconds. Sequential applications of up to 7 times per session are allowed for complete ablation of the lesions.

SUMMARY:
This study aims to evaluate the safety and efficacy of new ablation catheter developed by MEDICAL TAEWOONG for the treatment of pancreatic neoplasm (pancreatic adenocarcinoma or neuroendocrine tumour). The ablation is performed using EUSRA needle and radio frequency waves under ultrasound imaging. The subject who will be recruited into this study are patients who are deemed as non-surgical candidates.

DETAILED DESCRIPTION:
RFA causes tissue destruction through the application of a high frequency alternating current, generating local temperatures above 60°C and leading to coagulative necrosis. The technique has been widely used in many solid organ tumours and has been shown to result in 5-year survival rates comparable to surgery. The technique is currently the standard therapy in hepatocellular carcinoma and colorectal pulmonary metastasis particular in patients that are not suitable for surgery.

The application of RFA in the pancreas was first described in 1999. Thereafter, several studies performed in the porcine model demonstrated the feasibility of RFA under EUS guidance. In the first porcine study by Goldberg et al, RFA was applied through a modified 19 gauge Vilmann-type needle (GIP/MediGlobe, Grassau, Germany). The needles were electrically insulated with shrink tubing for all but the distal 1 to 1.5cm. 16 ablations were performed and the procedure resulted in hypodense foci of non-enhancing pancreas 1 to 2 days after ablation. Pathologic examination showed well demarcated spherical foci of coagulation necrosis measuring 8 to 12mm in size. One swine developed hyperlipasemia, a focal zone of pancreatitis and another with pancreatic fluid collection. 4 swine also suffered from thermal injury to the gastrointestinal wall caused by improper electrode placement.

Thereafter, 4 subsequent porcine studies also demonstrated the feasibility of RFA under EUS guidance with proprietary radiofrequency electrodes. In the most recent study, EUS-guided RFA was delivered by a novel 18-gauge RFA electrode and a VIVA RF generator (STARmed, Korea). RFA was applied to both the ex-vivo and in-vivo models to determine the optimum power settings and efficacy of the device. A power setting of 50 W for 6 minutes was shown to result in the most effective depth and size of ablation zone, whilst a higher power setting resulted in tissue charring and reduced the conductive coagulative necrosis effect. 10 swine then received EUS-guided RFA to the pancreas and the mean size of the ablated lesions were 23 +/- 6.9mm. None of the swine suffered from any adverse events and there were no significant changes in the serum levels of amylase and lipase, both before and after the procedures.

On the other hand, the experience of RFA in human pancreas is accumulating. Earlier studies using first generation percutaneous RFA probes applied intra-operatively to pancreatic carcinomas were associated with unacceptably high rates of mortality (0% - 25%) and morbidity (0% - 40%). Subsequently, human data on new generation EUS-guided RFA probes with improved design and outcomes have become available. 22 patients with locally advanced pancreatic ductal adenocarcinoma were treated the cryotherm probe (CTP) (ERBE Elektromedizin GmbH, Tübingen, Germany). The CTP was successfully applied in 16 patients (72.8%), amylase rose in 3 of 16 patients but none had clinical signs of pancreatitis. The median post ablation survival time was 6 months. In another 2 studies, the Habib RFA catheter was used (EMcision, United Kingdom). 7 patients with unresectable pancreatic ductal carcinoma and 8 patients with pancreatic neuroendocrine tumour and cystic tumours were treated with EUS-guided RFA. In patients suffering from pancreatic ductal carcinoma, post procedural imaging showed a decrease in size of the lesions in 2 patients and 1 patient suffered from mild pancreatitis. Whilst in patients with cystic neoplasms and neuroendocrine tumours, all showed complete resolution or reduction in size of the lesions. Only 2 patients suffered from abdominal pain that resolved spontaneously. On the other hand, RFA with the VIVA generator was applied in 6 patients with unresectable pancreatic adenocarcinoma. Two patients suffered from mild abdominal pain but no serious adverse events reported.

Thus, based on these preliminary results, we conclude that the new generation EUS-guided RFA probe is safe and feasible. The next stage in development with conduction of this study would involve recruitment of larger patient cohorts to further establish the efficacy and risk profile of the procedure.

HYPOTHESIS AND OBJECTIVES The aim of the current study is to perform a single center prospective study on EUS-guided radiofrequency ablation (RFA) of solid pancreatic neoplasms. We hypothesize that EUS-guided RFA is safe, feasible and effective for treating solid pancreatic neoplasms.

EXPECTED RIKS AND BENEFITS The expected risks for the patients include mild abdominal pain. The benefit may include RFA destroy the tumour cells via coagulative necrosis process hence providing some form of disease control. Besides, the current study could establish the safety and feasibility of EUS-guided RFA of solid pancreatic neoplasms. These results could provide insights as to whether the procedure is comparable to surgery for treatment of these lesions in the future.

STUDY POPULATION We aim to recruit 10 subjects over the period of 18 months. The subjects must have pancreatic neuroendocrine tumour or pancreatic ductal carcinoma that was unsuitable for surgery or not keen for surgery.

STUDY DESIGN AND PROCEDURES/METHODOLOGY The RFA system It consists of two components, a19-gauge RFA electrode and a VIVA combo RF generator. The total length of the electrode including the delivery system is 150 cm. The distal end of the electrode is needle-shaped and echogenic that allows EUS guided puncture of the target lesion. The active electrode tip is 1 cm in length. During ablation, the RF electrode is cooled and perfused internally with circulating chilled saline solution (0°C) delivered via a pump to maintain a constant temperature. A setting of 50W energy would be used for RFA and the duration of application is 10 seconds.

EUS-guided radiofrequency ablation This procedure is very similar to the standard technique of EUS-guided fine needle aspiration. The location and size of the lesion would be assessed for suitability of treatment. After locating the lesion, the RFA needle would be inserted to the centre of the lesion. RFA would then be initiated and hyperechoic interferences would be observed around the electrode signifying heating of the tissue. Post procedural, the site of needle entry would be inspected endoscopically to assess for presence of thermal injury to the gastrointestinal wall.

Follow-up protocol There will be clinic visit scheduled by both gastroenterologist and oncologist at two weeks after discharging from hospital to review participant's condition and to plan for further treatment. Follow-up phone call will be made at 1st week and 1st month after discharging from the ward to determine for any adverse event and whether they are attributable. When reporting complication rates, only definite and probably attributable events occurring within 30 days will be include.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years-old or above
* Suffering from pancreatic neuroendocrine tumour or pancreatic ductal carcinoma that was confirmed by fine needle aspiration cytology
* Unsuitable for surgery, due to one (or more) of the following items:

  * ASA score >/= III
  * An alternative advanced malignancy
  * Unsuitable for surgery upon expert's opinion for any other reason
* Individuals who are not keen for surgical resection
* Eligible for endoscopic intervention
* Written informed consent

Exclusion Criteria:

* Coagulopathy (international normalized ratio >1.5, partial thromboplastin time greater than twice that of control), platelet count <50,000x103/uL
* Pregnancy
* Patients with a poor mental condition or mental retardation, unable to understand the nature and possible consequences of the study
* Patients unwilling to undergo follow-up assessments
* Patients with liver cirrhosis, portal hypertension and/or gastric varices.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
To measure the technical success of EUS-guided RFA | 18 months
  It is defined as successful puncture of the pancreatic lesion with the RFA needle and completion of the ablation cycle.
To measure side effects and adverse event of EUS-guided RFA | 18 months
  Adverse events specific to RFA would be graded according to the lexicon of endoscopic adverse events (PB Cotton GIE 2010). Potential adverse events specific to RFA include:
  * Post-RFA syndrome: Combination of flu like symptoms including fever, malaise, pain at the site of ablation, nausea, and/or vomiting and that no other septic source is identified.
  * Pancreatitis: Clinical presence of abdominal pain with an increase in amylase level >3 times above the normal serum amylase levels.
  * Pancreatic leak: The presence of an abdominal collection with an amylase level that is >3 times normal serum amylase levels.
  * Thermal injury: Coagulative necrosis occurring at the site of needle entry within the gastrointestinal tract with or without clinical sequelae.

CONTACTS AND LOCATIONS:
Overall Officials: Yung Ka Chin, MBChB, Principal Investigator — Department of Gastroenterology & Herpetology, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD on study protocol will be made available
Supporting Information: Study Protocol
Time Frame: 12months after completion
Access Criteria: Information will be made available after requestors sign a data assess agreement.

REFERENCES:
- [Background] Rossi S, Fornari F, Pathies C, Buscarini L. Thermal lesions induced by 480 KHz localized current field in guinea pig and pig liver. Tumori. 1990 Feb 28;76(1):54-7. doi: 10.1177/030089169007600114. PMID 2181746
- [Background] McGahan JP, Browning PD, Brock JM, Tesluk H. Hepatic ablation using radiofrequency electrocautery. Invest Radiol. 1990 Mar;25(3):267-70. doi: 10.1097/00004424-199003000-00011. No abstract available. PMID 2185179
- [Background] Bai H, Huangz X, Jing L, Zeng Q, Han L. The effect of radiofrequency ablation vs. liver resection on survival outcome of colorectal liver metastases (CRLM): a meta-analysis. Hepatogastroenterology. 2015 Mar-Apr;62(138):373-7. PMID 25916066
- [Background] Qi X, Tang Y, An D, Bai M, Shi X, Wang J, Han G, Fan D. Radiofrequency ablation versus hepatic resection for small hepatocellular carcinoma: a meta-analysis of randomized controlled trials. J Clin Gastroenterol. 2014 May-Jun;48(5):450-7. doi: 10.1097/MCG.0000000000000008. PMID 24172183
- [Background] De Filippo M, Bozzetti F, Martora R, Zagaria R, Ferretti S, Macarini L, Brunese L, Rotondo A, Rossi C. Radiofrequency thermal ablation of renal tumors. Radiol Med. 2014 Jul;119(7):499-511. doi: 10.1007/s11547-014-0412-1. Epub 2014 Jul 15. PMID 25024061
- [Background] Smith SL, Jennings PE. Lung radiofrequency and microwave ablation: a review of indications, techniques and post-procedural imaging appearances. Br J Radiol. 2015 Feb;88(1046):20140598. doi: 10.1259/bjr.20140598. Epub 2014 Dec 3. PMID 25465192
- [Background] Liu SY, Ng EK, Lee PS, Wong SK, Chiu PW, Mui WL, So WY, Chow FC. Radiofrequency ablation for benign aldosterone-producing adenoma: a scarless technique to an old disease. Ann Surg. 2010 Dec;252(6):1058-64. doi: 10.1097/SLA.0b013e318f66936. PMID 21107117
- [Background] Keane MG, Bramis K, Pereira SP, Fusai GK. Systematic review of novel ablative methods in locally advanced pancreatic cancer. World J Gastroenterol. 2014 Mar 7;20(9):2267-78. doi: 10.3748/wjg.v20.i9.2267. PMID 24605026
- [Background] Kim HJ, Seo DW, Hassanuddin A, Kim SH, Chae HJ, Jang JW, Park DH, Lee SS, Lee SK, Kim MH. EUS-guided radiofrequency ablation of the porcine pancreas. Gastrointest Endosc. 2012 Nov;76(5):1039-43. doi: 10.1016/j.gie.2012.07.015. PMID 23078928
- [Background] Song TJ, Seo DW, Lakhtakia S, Reddy N, Oh DW, Park DH, Lee SS, Lee SK, Kim MH. Initial experience of EUS-guided radiofrequency ablation of unresectable pancreatic cancer. Gastrointest Endosc. 2016 Feb;83(2):440-3. doi: 10.1016/j.gie.2015.08.048. Epub 2015 Sep 4. PMID 26344883
- [Background] Chu KF, Dupuy DE. Thermal ablation of tumours: biological mechanisms and advances in therapy. Nat Rev Cancer. 2014 Mar;14(3):199-208. doi: 10.1038/nrc3672. PMID 24561446
- [Background] Goldberg SN, Mallery S, Gazelle GS, Brugge WR. EUS-guided radiofrequency ablation in the pancreas: results in a porcine model. Gastrointest Endosc. 1999 Sep;50(3):392-401. doi: 10.1053/ge.1999.v50.98847. PMID 10462663
- [Background] Varadarajulu S, Jhala NC, Drelichman ER. EUS-guided radiofrequency ablation with a prototype electrode array system in an animal model (with video). Gastrointest Endosc. 2009 Aug;70(2):372-6. doi: 10.1016/j.gie.2009.03.008. Epub 2009 Jun 26. PMID 19560138
- [Background] Carrara S, Arcidiacono PG, Albarello L, Addis A, Enderle MD, Boemo C, Campagnol M, Ambrosi A, Doglioni C, Testoni PA. Endoscopic ultrasound-guided application of a new hybrid cryotherm probe in porcine pancreas: a preliminary study. Endoscopy. 2008 Apr;40(4):321-6. doi: 10.1055/s-2007-995595. PMID 18389449
- [Background] Carrara S, Arcidiacono PG, Albarello L, Addis A, Enderle MD, Boemo C, Neugebauer A, Campagnol M, Doglioni C, Testoni PA. Endoscopic ultrasound-guided application of a new internally gas-cooled radiofrequency ablation probe in the liver and spleen of an animal model: a preliminary study. Endoscopy. 2008 Sep;40(9):759-63. doi: 10.1055/s-2008-1077520. Epub 2008 Aug 13. PMID 18702032
- [Background] Matsui Y, Nakagawa A, Kamiyama Y, Yamamoto K, Kubo N, Nakase Y. Selective thermocoagulation of unresectable pancreatic cancers by using radiofrequency capacitive heating. Pancreas. 2000 Jan;20(1):14-20. doi: 10.1097/00006676-200001000-00002. PMID 10630378
- [Background] Elias D, Baton O, Sideris L, Lasser P, Pocard M. Necrotizing pancreatitis after radiofrequency destruction of pancreatic tumours. Eur J Surg Oncol. 2004 Feb;30(1):85-7. doi: 10.1016/j.ejso.2003.10.013. PMID 14736529
- [Background] Hadjicostas P, Malakounides N, Varianos C, Kitiris E, Lerni F, Symeonides P. Radiofrequency ablation in pancreatic cancer. HPB (Oxford). 2006;8(1):61-4. doi: 10.1080/13651820500466673. PMID 18333241
- [Background] Wu Y, Tang Z, Fang H, Gao S, Chen J, Wang Y, Yan H. High operative risk of cool-tip radiofrequency ablation for unresectable pancreatic head cancer. J Surg Oncol. 2006 Oct 1;94(5):392-5. doi: 10.1002/jso.20580. PMID 16967436
- [Background] Spiliotis JD, Datsis AC, Michalopoulos NV, Kekelos SP, Vaxevanidou A, Rogdakis AG, Christopoulou AN. Radiofrequency ablation combined with palliative surgery may prolong survival of patients with advanced cancer of the pancreas. Langenbecks Arch Surg. 2007 Jan;392(1):55-60. doi: 10.1007/s00423-006-0098-5. Epub 2006 Nov 7. PMID 17089173
- [Background] Girelli R, Frigerio I, Salvia R, Barbi E, Tinazzi Martini P, Bassi C. Feasibility and safety of radiofrequency ablation for locally advanced pancreatic cancer. Br J Surg. 2010 Feb;97(2):220-5. doi: 10.1002/bjs.6800. PMID 20069610
- [Background] Arcidiacono PG, Carrara S, Reni M, Petrone MC, Cappio S, Balzano G, Boemo C, Cereda S, Nicoletti R, Enderle MD, Neugebauer A, von Renteln D, Eickhoff A, Testoni PA. Feasibility and safety of EUS-guided cryothermal ablation in patients with locally advanced pancreatic cancer. Gastrointest Endosc. 2012 Dec;76(6):1142-51. doi: 10.1016/j.gie.2012.08.006. Epub 2012 Sep 26. PMID 23021160
- [Background] 1. Pai M, Yang J, Zhang X, Jin Z, Wang D, Senturk H, Lakhtakia S, Reddy DN, Kahaleh M, Habib N, et al. Endoscopic ultrasound guided radiofrequency ablation (EUS-RFA) for pancreatic ductal adenocarcinoma. Gut. 2013;62(Suppl 1):A153.
- [Background] Pai M, Senturk H, Lakhtakia S, Reddy DN, Cicinnati C, Kabar I, Beckebaum S, Jin Z, Wang D, Yang J, et al. Endoscopic Ultrasound Guided Radiofrequency Ablation (EUS-RFA) for Cystic Neoplasms and Neuroendocrine Tumours of the Pancreas. Gastrointest Endosc. 2013;77(5S): AB143-AB144
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503